CLINICAL TRIAL: NCT02880787
Title: Comparison of Two Neuromuscular Transmission Monitors Based on Acceleromyography: TOF-Watch SX® and TOFScan®
Acronym: TOFScan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-A00540-47
Record Dates: First submitted 2016-08-18; First posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Curarisation; Neuromuscular Monitoring
MeSH Terms: interventions — Rocuronium; Neuromuscular Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Adult population 1 (Other): TOF-Watch SX® on nondominant arm and TOFScan® on dominant arm
  Interventions: Drug: Rocuronium; Device: Neuromuscular monitoring with TOFScan® and TOF-Watch SX®
- Adult population 2 (Other): TOF-Watch SX® on dominant arm and TOFScan® on nondominant arm
  Interventions: Drug: Rocuronium; Device: Neuromuscular monitoring with TOFScan® and TOF-Watch SX®
- Pediatric population 1 (Other): TOF-Watch SX® on nondominant arm and TOFScan® on dominant arm
  Interventions: Drug: Rocuronium; Device: Neuromuscular monitoring with TOFScan® and TOF-Watch SX®
- Pediatric population 2 (Other): TOF-Watch SX® on dominant arm and TOFScan® on nondominant arm
  Interventions: Drug: Rocuronium; Device: Neuromuscular monitoring with TOFScan® and TOF-Watch SX®

INTERVENTIONS:
Drug: Rocuronium — Anesthesia induction with Propofol and maintaining with desflurane. For adult patients, the curare is rocuronium (0.6 mg/kg) For pediatric patients, the curare can be rocuronium (0.6 mg/kg), cisatracurium (0.1 mg/kg) or atracurium (0.5 mg/kg)
Device: Neuromuscular monitoring with TOFScan® and TOF-Watch SX® — Each monitor on one arm

SUMMARY:
The purpose is to evaluate the reproducibility of neuromuscular monitoring data of recovery from neuromuscular blockade, obtained with TOFScan® and TOF-Watch SX®, in adult and pediatric population.

Secondary purposes are to evaluate the reproducibility of data obtained with 2 monitors for:

* the onset of clinical action of curare: suppression of the first response of train of four monitoring (T1) of 95% initial value
* the duration of clinical action of curare: recovery of the first response of train of four monitoring (T1) to 25% initial value
* recovery of first (T1), second (T2), third (T3) and fourth response (T4) of train of four monitoring, and recovery of T4/T1 to 40% and 60% initial value (T4/T1 0.4 and 0.6)
* complete recovery from curarisation, at T4/T1=90% and T4/T1=100%.

ELIGIBILITY:
Inclusion Criteria:

Adult population:

* Non opposition to research
* > 18 years old
* ASA score 1-3
* Undergoing surgery with curarisation through tracheal intubation
* Affiliation to social security

Pediatric population:

* > 1 year old
* Non opposition to research of child (if able to consent) or representatives with parental authority
* ASA score 1-4
* Undergoing surgery with curarisation
* Affiliation to social security

Exclusion Criteria:

Adult population:

* Allergy to administered drugs
* Known or suspected difficult intubation
* Pregnant women
* BMI > 40

Pediatric population:

* Allergy to administered drugs
* Known or suspected difficult intubation

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Time of recovery of the first (T1) response of train of four monitoring displayed on TOFScan and on TOF Watch SX | day 0, after induction of anesthesia
Time of recovery of the second (T2) response of train of four monitoring displayed on TOFScan and on TOF Watch SX | day 0, after induction of anesthesia
Time of recovery of the third (T3) response of train of four monitoring displayed on TOFScan and on TOF Watch SX | day 0, after induction of anesthesia
Time of recovery of the fourth (T4) response of train of four monitoring displayed on TOFScan and on TOF Watch SX | day 0, after induction of anesthesia
Time of recovery of T4/T1 of train of four monitoring at 40% of initial value displayed on TOFScan and on TOF Watch SX | day 0, after induction of anesthesia
Time of recovery of T4/T1 of train of four monitoring at 60% of initial value displayed on TOFScan and on TOF Watch SX | day 0, after induction of anesthesia
Time of recovery of T4/T1 of train of four monitoring at 90% of initial value displayed on TOFScan and on TOF Watch SX | day 0, after induction of anesthesia
Time of recovery of T4/T1 of train of four monitoring at 100% of initial value displayed on TOFScan and on TOF Watch SX | day 0, after induction of anesthesia

SECONDARY OUTCOMES:
Time of suppression of the first response of train of four monitoring (T1) at 95% initial value displayed on TOFScan and on TOF Watch SX | day 0, after induction of anesthesia
Time of recovery of the first response of train of four monitoring (T1) to 25% initial value displayed on TOFScan and on TOF Watch SX | day 0, after induction of anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Thomas FUCHS-BUDER, Pr, Principal Investigator — CHRU de NANCY - Hôpitaux de Brabois - Département d'Anesthésie-Réanimation - VANDOEUVRE LES NANCY - FRANCE
Locations (1):
- CHRU de NANCY - Hôpitaux de Brabois - Département d'Anesthésie-Réanimation, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No